CLINICAL TRIAL: NCT02999009
Title: A Prospective, Post-market, Multi-center Study of the Trident II Tritanium Acetabular Shell
Brief Title: Trident II Tritanium Acetabular Shell Outcomes Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 78
Record Dates: First submitted 2016-12-12; First posted 2016-12-21 (Estimated); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Arthroplasty, Replacement, Hip

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Trident II Tritanium Acetabular Shell (Other): The Trident II Tritanium Acetabular Shell is a hemispherical acetabular shell intended for use in a cementless application.
  Interventions: Device: Trident II Tritanium Acetabular Shell

INTERVENTIONS:
Device: Trident II Tritanium Acetabular Shell — A hemispherical acetabular shell indicated for cementless application.

SUMMARY:
The purpose of this study is to review the performance and success rate of an FDA approved cementless hip replacement part called the Trident II Tritanium Acetabular Shell. The study will specifically look at the need to revise the hip replacement after 5 years. This will be compared to how much this happens in patients who have hip replacement with similar cementless acetabular shells.

DETAILED DESCRIPTION:
This study is a prospective, open-label, post-market, non-randomized evaluation of the Trident II Tritanium Acetabular Shell for primary total hip arthroplasty (THA) with a cementless application in a consecutive series of patients who meet the eligibility criteria.

ELIGIBILITY:
Inclusion Criteria:

A. Patient has signed an Institutional Review Board (IRB) approved, study specific Informed Patient Consent Form.

B. Patient is a male or non-pregnant female age 18-80 years of age at the time of study device implantation.

C. Patient has primary diagnosis of Non-Inflammatory Degenerative Joint Disease.

D. Patient is a candidate for a primary cementless total hip replacement.

E. Patient is willing and able to comply with postoperative scheduled clinical and radiographic evaluations.

Exclusion Criteria:

F. Patient has a Body Mass Index (BMI) ≥ 40.

G. Patient is diagnosed with Inflammatory Arthritis.

H. Patient has an active or suspected latent infection in or about the affected hip joint at time of study device implantation.

I. Patient has a neuromuscular or neurosensory deficiency, which limits the ability to evaluate the safety and efficacy of the device.

J. Patient is diagnosed with a systemic disease (e.g. Lupus Erythematosus) or a metabolic disorder (e.g. Paget's Disease) leading to progressive bone deterioration.

K. Patient is immunologically suppressed or receiving steroids in excess of normal physiological requirements (e.g. > 30 days).

L. Patient requires revision surgery of a previously implanted total hip replacement or hip fusion to the affected joint.

M. Patient has had previous open surgery to the affected joint, not including arthroscopy.

N. Patient requires implantation of a constrained liner.

O. Patient has a known sensitivity to device materials.

P. Patient is a prisoner.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 383 (Actual)
Dates: Start 2017-01-20 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
Absence of Revision for the Trident II Tritanium Acetabular Shell | 5 years
  To demonstrate that acetabular replacement with the Trident II Tritanium Acetabular Shell provides clinical results comparable to similar acetabular components.

SECONDARY OUTCOMES:
All-cause Revision and Removal Rates for the Trident II Tritanium Acetabular Shell | 10 years
  Survivorship percentage (one reported value) for both all-cause revision + removal will be indicated
Radiographic Stability | 6 weeks, 3-6 months, 1, 2, 5, 7, 10 years
  Numerous parameters will be reviewed by zone, including radiolucency and migration.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Barga, Study Director — Director, Clinical Research - Stryker Joint Replacement
Locations (9):
- United States (9):
  - Tucson Orthopaedic Institute, Tucson, Arizona
  - Southeast Orthopedic Specialists, Jacksonville, Florida
  - American Hip Institute, Des Plaines, Illinois
  - Center for Orthopaedics and Spine, LLC, Lake Charles, Louisiana
  - St. Joseph Mercy Hospital Health System, Ypsilanti, Michigan
  - Rothman Institute, Egg Harbor, New Jersey
  - Hospital for Special Surgery, New York, New York
  - Northwell Health, Lenox Hill Hospital, New York, New York
  - UNC Orthopaedics, Chapel Hill, North Carolina